CLINICAL TRIAL: NCT00876252
Title: A Phase 2 Pilot Study Assessing Immunogenicity and Safety of IC43 in Intensive Care Patients
Brief Title: Study Assessing Immunogenicity and Safety of IC43 In Intensive Care Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IC43-201
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-10

CONDITIONS: Pneumonia, Ventilator-Associated
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- IC43 100 mcg (Active Comparator): IC43 100 mcg with Aluminum hydroxide
  Interventions: Biological: IC43
- IC43 200 mcg (Active Comparator): IC43 200 mcg with Aluminum hydroxide
  Interventions: Biological: IC43
- IC43 100 mcg w/o (Active Comparator): IC43 100 mcg without Aluminum hydroxide
  Interventions: Biological: IC43
- Placebo (Placebo Comparator): phosphate-buffered saline solution containing 0,9 % NaCl and 400 mcg Aluminum hydroxide as an adjuvant
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: IC43
  Other Names: IC43 Pseudomonas Aeruginosa
  Arms: IC43 100 mcg; IC43 100 mcg w/o; IC43 200 mcg
Drug: Placebo — NaCl
  Other Names: phosphate buffered saline (PBS)
  Arms: Placebo

SUMMARY:
Randomized, placebo-controlled, partially blinded phase 2 pilot study. Multicenter study (approximately 50 centers) in approximately 9 countries. Proposed start date is December 2008. The study duration per patient is estimated to be 90 days. Overall study duration is estimated to be 12-18 months.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, multi-center, partially blinded [i.e., 100 mcg and 200 mcg IC43 with Al(OH)3,, respectively] and placebo, but unblinded for non-adjuvanted IC43 [i.e., 100 mcg w/o Al(OH)3] phase 2 pilot study. The study population consists of male or female ICU patients with a need for mechanical ventilation for more than 48 hours, aged between 18 and 80 years.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients aged between 18 and 80 years
* Patients admitted to an ICU with a need for mechanical ventilation for more than 48 hours at visit 0
* At high risk for acquiring infection against P. aeruginosa at visit 0.
* Patients who, as determined by the investigator, have a high probability of survival for at least 48 hours.
* In females, either childbearing potential terminated by surgery or 1 year post menopausal, or a negative pregnancy test and the willingness of practicing a reliable methods of contraception
* Written informed consent or waiver according to the national regulations

Exclusion Criteria:

* Known use of any other investigational or non-registered drug within 30 days prior to IC43 vaccination at Visit 0
* Low severity of illness defined by an acute physiology score < 8 at visit 0
* Patients < 6 months post organ transplantation
* Severe thrombocytopenia or other coagulopathy which in the opinion of the investigator makes the patient unsuitable for intramuscular injection
* Pregnancy, lactation
* Persons who have been committed involuntarily to an institution, e.g. mental health facility or prison, will not participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Actual)
Dates: Start 2008-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

PRIMARY OUTCOMES:
Immunogenicity at day 14 as determined by OprF/I specific IgG antibody titer measured by ELISA in patients receiving IC43 or placebo | Day 14

SECONDARY OUTCOMES:
Immunogenicity at day 7 | Day 7
Rate of serious adverse events | Day 7
Safety laboratory parameters | Day 7
Systemic tolerability | Day 7
Local tolerability | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Haas, Study Director — Valneva Austria GmbH
Locations (1):
- Medical University of Vienna, Vienna, Vienna, Austria

REFERENCES:
- [Derived] Rello J, Krenn CG, Locker G, Pilger E, Madl C, Balica L, Dugernier T, Laterre PF, Spapen H, Depuydt P, Vincent JL, Bogar L, Szabo Z, Volgyes B, Manez R, Cakar N, Ramazanoglu A, Topeli A, Mastruzzo MA, Jasovich A, Remolif CG, Del Carmen Soria L, Andresen Hernandez MA, Ruiz Balart C, Kremer I, Molnar Z, von Sonnenburg F, Lyons A, Joannidis M, Burgmann H, Welte T, Klingler A, Hochreiter R, Westritschnig K. A randomized placebo-controlled phase II study of a Pseudomonas vaccine in ventilated ICU patients. Crit Care. 2017 Feb 4;21(1):22. doi: 10.1186/s13054-017-1601-9. PMID 28159015